CLINICAL TRIAL: NCT05752513
Title: Early vs Late Bladder Dissection During Cesarean Hysterectomy in Patients With Placenta Accreta Spectrum With Bladder Invasion
Brief Title: Early vs Late Bladder Dissection During CS Hysterectomy in Patients With PAS With Bladder Invasion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdalla Mousa, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-345-2022
Record Dates: First submitted 2023-02-22; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Placenta Accreta Spectrum; Cesarean Hysterectomy
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): 18 pregnant women scheduled for classical cesarean hysterectomy for placenta accreta
  Interventions: Procedure: early bladder dissection
- Group 2 (Experimental): 18 pregnant women scheduled for bladder last cesarean hysterectomy
  Interventions: Procedure: Late bladder dissection

INTERVENTIONS:
Procedure: Late bladder dissection — The bladder dissection is reserved as the last step of the cesarean hysterectomy with excellent dissection of the ureteric course till the ureteric tunnel to reduce the incidence of inadvertent ureteric clamping during uterine vessel ligating and transection
  Arms: Group 2
Procedure: early bladder dissection — The bladder dissection is early as in classic cesarean hysterectomy
  Arms: Group 1

SUMMARY:
Thirty-six singleton pregnant women with PAS and bladder invasion; total anterior or anterolateral invasion, who were scheduled for cesarean hysterectomy were randomly assigned into two equal groups

* Group 1: included 18 pregnant women scheduled for classical cesarean hysterectomy for placenta accreta with or without ligation of anterior division of internal iliac artery before cesarean section.
* Group 2: included 18 pregnant women scheduled for bladder last cesarean hysterectomy with or without ligation of anterior division of internal iliac artery.

ELIGIBILITY:
Inclusion Criteria:

1. Age: reproductive age.
2. Pregnant with singleton living fetus.
3. Previous one or more cesarean sections.
4. Gestational age: > 34 weeks.
5. Elective or non-emergency cesarean sections.
6. Preoperative hemoglobin more than 9.5 gm/dl.

Exclusion Criteria:

Women with history of any medical disorder with pregnancy eg. gestational diabetes, hypertension, or anemia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Amount of blood loss | during cesarean hysterectomy

SECONDARY OUTCOMES:
Operative time | during cesarean hysterectomy
bladder injury | during cesarean hysterectomy
ureteric injury | during cesarean hysterectomy
Need for massive blood transfusion | during cesarean hysterectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt